CLINICAL TRIAL: NCT02064309
Title: An Open Label, Pilot Investigation, to Assess the Safety and Efficacy of Transplantation of Macro-encapsulated Human Islets Within the Bioartificial Pancreas Beta-Air in Patients With Type 1 Diabetes Mellitus
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Beta-O2 Technologies Ltd. (Industry)
Responsible Party: Principal Investigator, Per-Ola Carlsson, Professor, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS Dnr2013/299
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Long-standing Type 1 Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human islets in Beta-Air device (Experimental)
  Interventions: Device: Beta-Air device for encapsulation of transplanted human islets

INTERVENTIONS:
Device: Beta-Air device for encapsulation of transplanted human islets

SUMMARY:
The primary objective of this clinical investigation is to investigate the safety of implantation of the human islet containing device Beta-Air in type 1 diabetic subjects.

The secondary objective of this clinical investigation is to investigate if the transplantation of macro-encapsulated human islets within the Beta-Air device can provide improved glycaemic control in type 1 diabetes patients with reduced incidences of hypoglycaemic episodes.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any investigation-related activities. Investigation-related activities are any procedure that would not have been performed during normal management of the subject.
2. Diagnosis of type 1 diabetes mellitus for > 5 years
3. Men or women > 18 years of age at the time of enrolment
4. Involvement in intensive diabetes management defined as self-monitoring of blood glucose level no less than a mean of three times per day averaged over each week and by the administration of three or more insulin injections per day or insulin pump therapy. This management must be under the direction of a diabetologist or diabetes specialist during the 12 months prior to study enrolment.

Exclusion Criteria:

1. Body mass index (BMI) > 30 kg/m²
2. Insulin requirement of > 1.0 Units/kg/day
3. HbA1c > 10 % (DCCT)
4. Random C-peptide > 0.003 nmol/l
5. Known untreated active proliferative diabetic retinopathy changes or increasing macular oedema
6. Renal failure (Glomerular Filtration Rate <60 ml/min)
7. Women of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or unwilling to use adequate contraceptive methods for the duration of the trial (implants, injectables, combined oral contraceptives, hormonal intrauterine device, sexual abstinence or vasectomised partner).
8. Active infection including hepatitis B, hepatitis C, HIV, Tbc
9. Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin
10. Known active alcohol or drug abuse.
11. Any coagulopathy or medical condition that would require long-term anticoagulant therapy (e.g., Warfarin) after transplantation (low-dose aspirin treatment is allowed) or subjects with an international normalized ratio (INR) > 1.5.
12. Severe co-existing cardiac disease, characterized by any of these conditions:

    1. Recent myocardial infarction (within past 36 weeks)
    2. Evidence of ischemia on functional cardiac exam within the last year
    3. Left ventricular ejection fraction < 30 %
    4. Cardiovascular conditions within 36 weeks prior to this trial:

    i. Decompensated heart failure New York Heart Association (NYHA) class III or IV ii. Unstable angina pectoris iii. Coronary arterial bypass graft iv. Coronary angioplasty
13. Inadequately treated blood pressure elevation (systolic BP > 160 mmHg or diastolic blood pressure > 100 mmHg)
14. Use of any medications to treat diabetes other than insulin within 4 weeks of enrolment
15. Administration of live attenuated vaccine(s) within 8 weeks of enrolment
16. Any previous organ transplant
17. Treatment with any immunosuppressive drug
18. Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial (e.g., systemic glucocorticoids)
19. Known or suspected allergy of hypersensitivity to trial product(s) or related products
20. The receipt of any investigational product within 30 days of screening for this trial
21. Any scheduled transplant in addition to the islet transplantation
22. Fulfillment of criteria for clinical pancreas or islet transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Safety of device, as evaluated by incidence of adverse events or serious adverse events judged probable or highly probable related to the device | 0-365 days

SECONDARY OUTCOMES:
1. Incidence of local or systemic inflammation or infection, incl. C-reactive protein rise, judged related to the device during course of study. | 0-365 days
2. Incidence and severity of fibrosis surrounding the device during course of study. | 0-365 days
3. Signs of immunization in transplanted patients. | 0-365 days
4. Oxygenation of tissue in the device, as evaluated at 4, 12 and 26 weeks post-transplantation | 0-180 days
5. Survival of endocrine tissue in the device, as evaluated by [11C]-5-hydroxytryptophane positron emission tomography and histological analysis at 26 weeks post-transplantation. | 0-180 days
6. Numbers of patients with peak c-peptide >0.20 nmol/l, in response to the mixed meal tolerance test at 12 and 26 weeks post-transplantation | 12 and 26 weeks post-transplantation
7. C-peptide area under the curve in response to the mixed meal tolerance test at 12 and 26 weeks post-transplantation. | 12 and 26 weeks post-transplantation
8. Number of patients with non-fasting c-peptide concentrations >0.003 nmol/l at 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 and 26 weeks post-transplantation; i.e. Kaplan-Meier analysis of survival time for islet grafts. | 0-26 weeks

OTHER OUTCOMES:
1. Number of patients with daily insulin needs <0.25 Units/kg at 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 and 26 weeks post-transplantation | 0-26 weeks post-transplantation
2. Delta changes in insulin requirement/kg body weight at 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 and 26 weeks post-transplantation when compared to before transplantation and 6 months after explantation | 0-365 days
3. Delta changes in glycosylated hemoglobin (HbA1c) at 2, 4, 8, 12, 14, 18 and 26 weeks post-transplantation when compared to before transplantation and 6 months after explantation. | 0-365 days
4. Delta changes in P-fructosamine at 2, 4, 8, 12, 18 and 26 weeks post-transplantation when compared to before transplantation and 6 months after explantation. | 0-365 days
5. Delta changes in glucose variability and hypo/hyper glycaemia duration derived from a continuous glucose monitoring system performed at 12 and 26 weeks post-transplantation when compared to before transplantation and 6 months after explantation. | 0-365 days
6. Quality of Life in transplanted patients at 12 and 26 weeks post-transplantation when compared to before transplantation and 6 months after explantation. | 0-365 days
7. Score in diabetes treatment satisfaction questionnaire in transplanted patients at 12 and 26 weeks post-transplantation when compared to before transplantation and 6 months after explantation. | 0-365 days

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Carlsson PO, Espes D, Sedigh A, Rotem A, Zimerman B, Grinberg H, Goldman T, Barkai U, Avni Y, Westermark GT, Carlbom L, Ahlstrom H, Eriksson O, Olerud J, Korsgren O. Transplantation of macroencapsulated human islets within the bioartificial pancreas betaAir to patients with type 1 diabetes mellitus. Am J Transplant. 2018 Jul;18(7):1735-1744. doi: 10.1111/ajt.14642. Epub 2018 Feb 2. PMID 29288549